CLINICAL TRIAL: NCT03665012
Title: The Pediatric Development Clinic Study: the Development, Medical and Nutritional Outcomes of Children Discharged From the Neonatal Unit in Rural Rwanda
Brief Title: The Pediatric Development Clinic Study
Acronym: PDC
Status: Completed | Type: Observational
Sponsor: Partners in Health (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Catherine Kirk, Director of Maternal and Child Health, Partners in Health
Other Study IDs: 222
Record Dates: First submitted 2017-10-11; First posted 2018-09-11 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Pregnancy, Puerperium and Perinatal Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pediatric Development Clinic (PDC) — All children enrolled in PDC will be at screened for any medical condition they may have and be referred for treatment as required. Nutrition and development support are also provided to clinic enrollees, based on clinic protocols which include regular monitoring and intervention.

SUMMARY:
Many preterm, low birth weight and other high-risk infants are surviving the early neonatal period. However, upon discharge from the neonatal units, this at-risk population has little support for their health, nutrition and development in the community. To address this emerging need, Partners In Health in collaboration with the Ministry of Health and UNICEF, has created a pediatric developmental clinic (PDC) to follow the high-risk infants after discharge from hospitals and health centers.

DETAILED DESCRIPTION:
Neonatal health and improving neonatal mortality has become one of the top priorities globally. In Rwanda, hospital care has advanced significantly with the development of national neonatal care guidelines and widespread provider training. As advances in technology and resuscitation become more commonly available, many preterm, low birth weight and other high-risk infants are surviving the early neonatal period. However, upon discharge from the neonatal units, this at-risk population has little support for their health, nutrition and development in the community. To address this emerging need, Partners In Health in collaboration with the Ministry of Health and UNICEF, has created a pediatric developmental clinic (PDC) to follow the high-risk infants after discharge from hospitals and health centers. Prior to implementation, a community-based descriptive study assessing the baseline medical, nutritional and developmental needs of low-birth weight and preterm infants who are the target population of the pediatric development clinic was conducted (Baseline Phase One). Subsequently, after 1-2 years of implementation an evaluation of clinical, nutritional and developmental outcomes of children followed in PDC will be conducted in comparison with the baseline study outcomes (Post-PDC Phase Two). Ongoing research on PDC implementation will focus on research on patient and provider experiences, overall clinic processes, cost-effectiveness, expansion of the PDC model, decentralization to health centers, and longer term outcomes of children enrolled in the PDC to further help refine the PDC model (Post-PDC Phase Three)

ELIGIBILITY:
Inclusion Criteria:

* All under-five children meeting PDC referral criteria as described in the study population description will be enrolled in PDC.

Exclusion Criteria:

* Patients who do not meet referral criterial for PDC or who are over age 5 years.

Ages: 1 Week to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All under-five children in need of formal follow-up with the following medical condition will be enrolled in PDC
  * children born premature
  * children born with an extremely low birth weight (ELBW)/ very low birth weight (VLBW)
  * infants born at term with HIE or Central Nervous System infections (cerebral malaria and meningitis)
  * children with developmental delays,
  * children with trisomy 21, hydrocephalus, cleft lip/palate
  * children less than 12 months of age discharged from the hospital following malnutrition treatment.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
To compare developmental outcomes of children who were enrolled in the PDC to children who did not receive PDC services and to the general population. | April 2014 to March 2019
  Proportion of children who are on track developmentally measured by the Ages and Stages Questionnaire Version 3 (ASQ-3) and Caregiver Reported Early Childhood Development Index (CREDI).

SECONDARY OUTCOMES:
To compare nutritional outcomes of children who were enrolled in the PDC to children who did not receive PDC services and to the general population. | April 2014 to March 2019
  Proportion of children with normal nutritional status based on anthropometric measures and World Health Organization Growth Standards: weight-for-age (underweight) or weight-for-height (wasting) or length/height-for-age (stunting) z-scores < -2 (undernutrition) vs healthy (z-score >-2).

CONTACTS AND LOCATIONS:
Locations (1):
- Kirehe District Hospital, Kirehe, Eastern, Rwanda

IPD SHARING:
Plan to Share IPD: No
Individual children data can only be shared on request according to the Rwandan policy on data sharing. However, study findings will be shared in different meetings, conferences and journals.

REFERENCES:
- [Result] Bayitondere S, Biziyaremye F, Kirk CM, Magge H, Hann K, Wilson K, Mutaganzwa C, Ngabireyimana E, Nkikabahizi F, Shema E, Tugizimana DB, Miller AC. Assessing retention in care after 12 months of the Pediatric Development Clinic implementation in rural Rwanda: a retrospective cohort study. BMC Pediatr. 2018 Feb 16;18(1):65. doi: 10.1186/s12887-018-1007-0. PMID 29452576
- [Result] Ngabireyimana E, Mutaganzwa C, Kirk CM, Miller AC, Wilson K, Dushimimana E, Bigirumwami O, Mukakabano ES, Nkikabahizi F, Magge H. A retrospective review of the Pediatric Development Clinic implementation: a model to improve medical, nutritional and developmental outcomes of at-risk under-five children in rural Rwanda. Matern Health Neonatol Perinatol. 2017 Jul 12;3:13. doi: 10.1186/s40748-017-0052-2. eCollection 2017. PMID 28706729
- [Derived] Nemerimana M, Karambizi AC, Umutoniwase S, Barnhart DA, Beck K, Bihibindi VK, Wilson K, Nshimyiryo A, Bradford J, Havugarurema S, Uwamahoro A, Nsabyamahoro E, Kirk CM. Evaluation of an mHealth tool to improve nutritional assessment among infants under 6 months in paediatric development clinics in rural Rwanda: Quasi-experimental study. Matern Child Nutr. 2021 Oct;17(4):e13201. doi: 10.1111/mcn.13201. Epub 2021 May 7. PMID 33960693

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03665012/Prot_SAP_000.pdf